CLINICAL TRIAL: NCT02476188
Title: Neutrophil Extracellular Traps and Thrombolysis in the Acute Stroke
Acronym: NETs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D15-P007
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Acute Stroke
Keywords: Neutrophil extracellular traps, stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients (Experimental): Samples of blood at H0, H+6, H+24 and H+72
  Interventions: Procedure: Sample of Blood
- Patients control (Experimental): Samples of blood at H0
  Interventions: Procedure: Sample of Blood
- Control (healthy person) (Active Comparator): Samples of blood at H0
  Interventions: Procedure: Sample of Blood

INTERVENTIONS:
Procedure: Sample of Blood

SUMMARY:
The purpose of the study was to investigate the correlation between the nucleosome concentration and the rate of recanalization after thrombolysis. All patients were admitted to the Stroke Unit at the University Hospital Sainte-Anne where they received standard stroke care. The investigators included all patients treated or not by intravenous thrombolysis for anterior circulation stroke with or without vessel occlusion. Exclusion criteria were neoplasms, chronic inflammatory diseases and cytostatic therapy at the time of stroke and stroke-specifics symptoms that had started earlier than 4.5 hours before admission.

DETAILED DESCRIPTION:
Neutrophil extracellular traps (NETs) were measured in serum at the time of hospitalization, then at 4 hours, 24 hours and 72 hours after stroke. Because of nucleosome instability, a strict preanalytical protocol was followed. Blood samples were centrifuged within 1-2 h after blood drawing. A strict preanalytical protocol was followed including early centrifugation of the samples and storage at - 80°C. NETs were quantified in batches containing all samples from a patient using the detection of MPO (myeloperoxidase) then the Cell-Death-Detection ELISAPLUS (Roche Diagnostics, Germany) as described earlier. Nucleosomes were quantified in relative arbitrary units (AU). Blood samples from each patient were measured within the same run to improve the comparability of the results.

For statistical analysis, various variables of nucleosomes were considered, such as the absolute concentrations determined at admission, at 24 hours and at 72 hours after stroke. Influence of nucleosome concentration on recanalization was tested. Continuous correlations of nucleosomes and infarction volume, nucleosomes and clot size, as well as of infarction volume and NIHSS were calculated by Spearman's rank correlation together with the 95% confidence interval. A p value < 0.05 was considered statistically significant.

The extent of the morphological damage was determined at time of admission to the hospital and 24 hours after thrombolysis by diffusion-weighted magnetic resonance imaging (MRI). The pretreat¬ment and follow-up DWI lesions was segmented using interactive tools based on DWI signal intensity thresholding within a 3-dimensional mask encompassing the apparent area of bright DWI signal intensity and morphometric filtering. The clot location and length were assessed on the susceptibility vessel sign on T2* as describe earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients ("Patients" + "Patients control" groups) :

Inclusion-1st sample of blood : every patient recruited within the neurovascular unit of intensive care of the Hospital center Sainte - Anne within the framework of a "thrombolyse alert ".

Then pursuit of the study ("patients" group only) if :

* Age 18 minimum
* Sylvien Infarct proved by the intellectual MRI,
* Whatever is the treatment received (Aspegic, thombolysis and/or thrombectomy)
* That there is occlusion of a cerebral artery or not "Controls" group :
* Healthy subjects,
* Mated on the age and the vascular risk factors (tobacco, arterial high blood pressure, diabetes and dyslipidémie)

Exclusion Criteria:

* Patients:
* Contraindications in the intravenous thrombolysis according to the current recommendations .

  * Controls:
* Histories of evolutionary pathology or thrombo-embolique, taken by treatment whatever it is except contraceptive for the women, the viral or bacterial infection in the month precedents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate of recanalisation | 24 hours
  Correlation between NETs and stroke severity

SECONDARY OUTCOMES:
Thrombus size on MRI | 24 hours
  Correlation between NETs and stroke severity
Stroke volume on MRI | 24 hours
  Correlation between NETs and stroke severity

CONTACTS AND LOCATIONS:
Overall Officials: Michel PLOTKINE, PhD, Study Director — University of Paris 5 - Rene Descartes
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France

REFERENCES:
- [Background] Holdenrieder S, Stieber P, Bodenmuller H, Fertig G, Furst H, Schmeller N, Untch M, Seidel D. Nucleosomes in serum as a marker for cell death. Clin Chem Lab Med. 2001 Jul;39(7):596-605. doi: 10.1515/CCLM.2001.095. PMID 11522104
- [Background] Holdenrieder S, Stieber P, Chan LY, Geiger S, Kremer A, Nagel D, Lo YM. Cell-free DNA in serum and plasma: comparison of ELISA and quantitative PCR. Clin Chem. 2005 Aug;51(8):1544-6. doi: 10.1373/clinchem.2005.049320. No abstract available. PMID 16040855
- [Background] Naggara O, Raymond J, Domingo Ayllon M, Al-Shareef F, Touze E, Chenoufi M, Gerber S, Mellerio C, Zuber M, Meder JF, Mas JL, Oppenheim C. T2* "susceptibility vessel sign" demonstrates clot location and length in acute ischemic stroke. PLoS One. 2013 Oct 11;8(10):e76727. doi: 10.1371/journal.pone.0076727. eCollection 2013. PMID 24146915